CLINICAL TRIAL: NCT01779440
Title: Decision Support for Smoking Cessation in Young Adults With Severe Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mary F. Brunette, MD, Associate Professor MD, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R21CA158863-01A1 (NIH); R21CA158863-01A1 (NIH)
Record Dates: First submitted 2013-01-25; First posted 2013-01-30 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-05

CONDITIONS: Mental Illness; Tobacco Smoking; Psychotic Disorders
Keywords: Mental Illness; Tobacco Smoking; Young Adults; Treatment Engagement; Motivational Intervention
MeSH Terms: conditions — Mental Disorders; Tobacco Smoking; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electronic Decision Support System (Other): The Electronic Decision Support System is a web-based computer program designed to motivate, educate, and engage people with severe mental illness into evidence-based smoking cessation treatment.
  Interventions: Behavioral: Electronic Decision Support System
- Control Computer Program (Placebo Comparator): A computer program aimed to educate people about smoking cessation treatment.
  Interventions: Behavioral: Electronic Decision Support System

INTERVENTIONS:
Behavioral: Electronic Decision Support System

SUMMARY:
Up to 77% of young people with severe mental illnesses smoke, a rate that is up to five times higher than the rate of daily smoking in other young adults. Contrary to popular belief, smoking tobacco does not provide any benefit for mental illness symptom control. People with severe mental illnesses (SMI: schizophrenia and severe mood disorders) are dying, on average, 25 years earlier than those without SMI. Much of this early mortality is due to higher rates of heart and lung diseases, cancers, strokes, and diabetes.

Cessation of smoking in these transition-age young adults can prevent cancer and increase life expectancy to that of non-smokers. Combination treatments are effective in this group and therefore key to improving outcomes, but few SMI smokers use them despite their interest in quitting. Motivational interventions for cessation increase interest in quitting, but public mental health clinicians do not deliver them, in part due to economic reasons. Thus cost effective methods to deliver motivational interventions to engage young smokers with SMI into treatment are needed.

To address this gap, we have developed an electronic decision support system (EDSS) for smoking cessation that is specifically tailored for smokers with SMI, who tend to have cognitive deficits and limited computer experience. Similar to EDSSs developed for other health problems, this EDSS provides information and motivational exercises within an easy-to-use, web-based computer program that can be used with minimal or no staff assistance. Initial piloting of the EDSS in middle-aged SMI smokers showed excellent usability and promising efficacy. Pilot-testing among young patients suggested that the EDSS increased motivation to quit smoking and provided direction to adapt the format and content of the EDSS for young SMI smokers.

The purpose of this proposal is to further develop the motivational decision support system and to test its ability to motivate young smokers with SMI to quit smoking with cessation treatment.

DETAILED DESCRIPTION:
The research will take place over 2 years at the Long Island Zucker Hillside Hospital system. In Year 1, we will adapt our electronic decision support system, a web-based motivational tool, for young smokers with severe mental illness. We will first identify beliefs of young smokers with severe mental illness that impede use of smoking cessation treatments. Then, the decision support system will be revised to change these beliefs, field-tested for usability, and improved as needed. In Year 2, we will conduct a randomized control trial of the newly revised version of the system among 60 young smokers with severe psychotic disorders.

In the controlled trial, participants will be assessed at baseline for mental health symptoms and smoking behavior and history, and then randomized to use the system or a computerized public health pamphlet (control condition) within two weeks. Participants will be assessed again at 14-week follow-up for clinician-confirmed initiation of smoking cessation treatment (main outcome), beliefs, and smoking characteristics. Analyses will assess whether use of the decision support system results in greater initiation of cessation treatment (main outcome), and changes in beliefs about treatment, than use of the control intervention.

ELIGIBILITY:
Inclusion Criteria:

English-speaking; non-pregnant/nursing; daily smokers; age 18-30; psychiatrically stable; in treatment in the Zucker Hillside Hospital system; diagnosed with SMI (schizophrenia, schizoaffective disorder, or mood disorder with psychotic features from medical chart); willing and able to give informed consent.

Exclusion Criteria:

(Phase 4 only): current (within the past month) use of evidence-based smoking cessation treatment (indicating the subject is already motivated), psychiatric instability (Modified Colorado Symptom Index score >45), current untreated substance use disorder (SUD)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2018-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary F. Brunette, MD, Principal Investigator — Dartmouth College
Locations (3):
- United States (3):
  - Mental Health Center of Greater Manchester, Manchester, New Hampshire
  - Greater Nashua Mental Health Center, Nashua, New Hampshire
  - Zucker-Hillside Hospital, Glen Oaks, New York

REFERENCES:
- [Background] Brunette MF, Feiron JC, Aschbrenner K, Colctti D, Devitt T, Greene MA, Harrington A, MoHugo GC, Pratt S, Robinson D, Williams J, Xie H. Characteristics and Predictors of Intention to use Cessation Treatment among Smokers with Schizophrenia: Young Adults Compared to Older Adults. J Subst Abus Alcohol. 2017;5(1):1055. Epub 2017 Mar 23. PMID 29881770
- [Result] Brunette MF, Ferron JC, Robinson D, Coletti D, Geiger P, Devitt T, Klodnick V, Gottlieb J, Xie H, Greene MA, Ziedonis D, Drake RE, McHugo GJ. Brief Web-Based Interventions for Young Adult Smokers With Severe Mental Illnesses: A Randomized, Controlled Pilot Study. Nicotine Tob Res. 2018 Sep 4;20(10):1206-1214. doi: 10.1093/ntr/ntx190. PMID 29059417

RESULTS

PARTICIPANT FLOW:
Groups:
- Electronic Decision Support System: The Electronic Decision Support System is a web-based computer program designed to motivate, educate, and engage people with severe mental illness into evidence-based smoking cessation treatment.
  Electronic Decision Support System
- Control Computer Program: A computer program aimed to educate people about smoking cessation treatment.
  Electronic Decision Support System
Period: Overall Study
Arm/Group | Electronic Decision Support System | Control Computer Program
Started | 30 | 28
Completed | 27 | 23
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Electronic Decision Support System | Control Computer Program | Total
Number analyzed (Participants) | 30 | 28 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.5 (3.9) | 25.0 (3.2) | 24.2 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 20 | 19 | 39
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 17 | 16 | 33
  African American | 9 | 10 | 19
  Other race | 4 | 2 | 6
Mean cigarettes per day [Mean (Standard Deviation); unit: cigarettes] | 10.9 (8.6) | 13.9 (9.4) | 12.3 (9.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Utilized Smoking Cessation Treatment
Description: Assesses through clinician confirmation any engagement in behavioral smoking cessation treatment and/or smoking cessation medication treatment.
Time Frame: 14 week follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Electronic Decision Support System | Control Computer Program
Number analyzed (Participants) | 27 | 23
Participants | 2 | 1
Statistical Analysis 1: Comparison: Electronic Decision Support System vs Control Computer Program; Test type: Superiority; p = 0.65, Chi-squared — The P-Value of 0.65 was calculated from the difference between groups for the above outcome variable

2. Secondary Outcome: Number of Participants With Biologically Confirmed Abstinence
Description: Abstinence - self report for past 7 days confirmed with breath Carbon Monoxide <9 ppm
Time Frame: 14 weeks
Population: Participants who attended the follow-up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Electronic Decision Support System | Control Computer Program
Number analyzed (Participants) | 27 | 23
Participants | 4 | 0

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | Electronic Decision Support System | Control Computer Program
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/28
Other Adverse Events (participants affected / at risk) | 0/30 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-11-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT01779440/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT01779440/SAP_001.pdf